CLINICAL TRIAL: NCT04740164
Title: A Randomized Study to Compare LMA® Gastro™, a Dual Channel Supraglottic Airway (SGA) Device, to Oxygenation With Standard Nasal Cannula for Endoscopic Retrograde Cholangiopancreatography (ERCP)
Brief Title: A Dual Channel Supraglottic Airway Device (LMA Gastro) for Oxygenation in Patients Undergoing ERCP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2020-1014; NCI-2021-00118 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2020-1014 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2021-01-29; First posted 2021-02-05 (Actual); Results first posted 2024-11-06 (Actual); Last update posted 2024-11-06 (Actual); Status verified 2024-11

CONDITIONS: Bile Duct Carcinoma; Gallbladder Carcinoma; Pancreatic Ductal Adenocarcinoma
MeSH Terms: conditions — Bile Duct Neoplasms; Gallbladder Neoplasms | interventions — Cholangiopancreatography, Endoscopic Retrograde

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Arm I (ERCP with LMA Gastro) (Experimental): Patients undergo ERCP with LMA Gastro.
  Interventions: Procedure: Endoscopic Retrograde Cholangiopancreatography
- Arm II (ERCP with standard nasal cannula) (Active Comparator): Patients undergo ERCP with standard nasal cannula.
  Interventions: Procedure: Endoscopic Retrograde Cholangiopancreatography

INTERVENTIONS:
Procedure: Endoscopic Retrograde Cholangiopancreatography — Undergo ERCP with LMA Gastro
  Other Names: ERCP
  Arms: Arm I (ERCP with LMA Gastro)
Procedure: Endoscopic Retrograde Cholangiopancreatography — Undergo ERCP with standard nasal cannula
  Other Names: ERCP
  Arms: Arm II (ERCP with standard nasal cannula)

SUMMARY:
This clinical trial compares the effect of LMA Gastro, a dual channel supraglottic airway (SGA) device, to oxygenation with standard nasal cannula for endoscopic retrograde cholangiopancreatography (ERCP). An ERCP is a combination of imaging scans and endoscopy that helps doctors diagnose and treat conditions of the pancreas and bile ducts that requires general anesthesia or procedural sedation. Anesthesiologists often use SGAs or nasal cannulas to help patients breathe while they are asleep during procedures. An SGA consists of an airway tube that connects to a mask, which is inserted through the mouth and placed at the back of the throat to keep the airway open while patients are under anesthesia or sedation. The nasal cannula is a device that fits in a patient's nostrils and delivers oxygen through a small, flexible tube while they are under anesthesia or sedation. The goal of this trial is to compare the effects of the LMA Gastro to nasal cannula when used to deliver oxygen to patients while they are asleep during their ERCP procedure.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To compare the incidence of desaturation (oxygen saturation [SpO2] < 90%) between patients undergoing ERCP with LMA Gastro versus (vs) standard nasal cannula.

SECONDARY OBJECTIVES:

I. To evaluate the incidence of additional airway maneuvers (jaw thrust/chin lift/placement of oral airway or/nasal trumpet/intubation).

II. To evaluate the incidence of withdrawal of duodenoscope from the airway to facilitate airway support.

III. To evaluate the incidence of adverse events. IV. To evaluate times related to anesthesia and procedure (defined as "anesthesia start to anesthesia end" and "procedure start to procedure end" respectively).

V. To evaluate time from procedure end to anesthesia end. VI. To describe hemodynamics within the two groups (recorded blood pressures, heart rates, oxygen saturations, and end tidal carbon dioxide [CO2]).

VII. To evaluate anesthesiologist placing the device (training video viewed, number of practice attempts, years of experience).

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM I: Patients undergo ERCP with LMA Gastro.

ARM II: Patients undergo ERCP with standard nasal cannula.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (>= 18 years old) undergoing ERCP

Exclusion Criteria:

* Patients with propofol allergy
* Patients at increased aspiration risk
* Patients with abnormal head/neck pathology preventing LMA Gastro placement
* Patients with surgical or radiation treatment to the head/neck making LMA Gastro placement difficult
* Patient with known difficult airway requiring advanced intubation equipment (with the exception of the video-laryngoscope) in the past
* Esophagectomy patients
* Patients already intubated upon arrival to endoscopy suite
* Patients undergoing endoscopic ultrasound (EUS)
* Patients with body mass index (BMI) >= 35 kg/m^2
* Patients with hypoxemia (SpO2 < 94% on room air or on home oxygen)
* American Society of Anesthesiology (ASA) Physical Status IV-V

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2021-02-24 (Actual); Primary Completion 2023-05-04 (Actual); Study Completion 2023-05-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Katherine Hagan, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: M D Anderson Cancer Center — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study enrolled 66 patients from 02/24/2021 to 06/24/2022. Patients ≥18 years old undergoing elective ERCP with TIVA were eligible for enrollment.
Groups:
- LMA Gastro: This group of patients received GA during their procedure, using LMA Gastro for intubation.
- Standard of Care: This group received TIVA during their procedure.
Period: Overall Study
Arm/Group | LMA Gastro | Standard of Care
Started | 33 | 33
Completed | 26 | 30
Not Completed | 7 | 3
Not completed — Lack of Efficacy | 4 | 0
Not completed — Physician Decision | 3 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | LMA Gastro | Standard of Care | Total
Number analyzed (Participants) | 26 | 30 | 56
Age, Continuous [Mean (Full Range); unit: years] | 56.6154 [23 to 77] | 62.8667 [42 to 85] | 59.96 [23 to 85]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 8 | 23
  Male | 11 | 22 | 33
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 26 | 30 | 56
ASA Status (grade) [Count of Participants; unit: Participants]
  II (better) | 0 | 1 | 1
  III (worse) | 26 | 29 | 55

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants That Had Desaturation Episodes of SpO2 <90%
Description: The desaturation (SpO2 < 90%) between patients undergoing ERCP with LMA® Gastro™ vs standard nasal cannula
Time Frame: The time between Anesthesia Start time and Anesthesia End time, 1.5 hrs in average
Measure: Count of Participants; unit: Participants
Arm/Group | LMA Gastro | Standard of Care
Number analyzed (Participants) | 26 | 30
Participants
  Desaturation <90% - Yes | 0 | 3
  Desaturation <90% - No | 26 | 27

2. Secondary Outcome: Incidence of Additional Airway Maneuvers
Description: Number of Participants that required additional manuevers to secure airway during their surgery
Time Frame: The time between Anesthesia Start time and Anesthesia End time, 1.5 hrs in average
Measure: Count of Participants; unit: Participants
Arm/Group | LMA Gastro | Standard of Care
Number analyzed (Participants) | 26 | 30
Participants
  Yes | 5 | 19
  No | 21 | 11

3. Secondary Outcome: Incidence of Withdrawal of Duodenoscope From Airway to Facilitate Airway Support
Description: Patients in which Duodenoscope was withdrawn to facilitate airway support
Time Frame: The time between Anesthesia Start time and Anesthesia End time
Measure: Count of Participants; unit: Participants
Arm/Group | LMA Gastro | Standard of Care
Number analyzed (Participants) | 26 | 30
Participants
  Yes | 9 | 10
  No | 17 | 20

4. Secondary Outcome: Incidence of Adverse Events
Description: Number of adverse events reported by the participants and/or reported by care providers during Surgery and in PACU, 3 hrs in average
Time Frame: From PACU arrival to PACU discharge, 3 hours in average
Measure: Number; unit: events
Arm/Group | LMA Gastro | Standard of Care
Number analyzed (Participants) | 26 | 30
events | 24 | 3

5. Secondary Outcome: To Evaluate Times Related to Anesthesia and Procedure
Description: Defined as "anesthesia start to anesthesia end" and "procedure start to procedure end" respectively
Time Frame: From anesthesia start to anesthesia end" and "procedure start to procedure end, up to 165 minutes
Measure: Mean (Full Range); unit: minutes
Arm/Group | LMA Gastro | Standard of Care
Number analyzed (Participants) | 26 | 30
minutes
  Total Anesthesia Time | 75.0769 [46 to 152] | 62.8667 [35 to 165]
  Total Procedure Time | 32.6154 [3 to 113] | 45.5333 [13 to 143]

6. Secondary Outcome: To Evaluate Time From Procedure End to Anesthesia End
Description: The time elapsed between procedure end and anesthesia end
Time Frame: From procedure end and anesthesia end, up to 60 minutes
Measure: Mean (Full Range); unit: minutes
Arm/Group | LMA Gastro | Standard of Care
Number analyzed (Participants) | 26 | 30
minutes | 18.5769 [10 to 49] | 11.2 [2 to 22]

7. Secondary Outcome: To Describe Heart Rates Within the Two Groups
Description: Heart rates were measured prior treatment administration and at the end of the procedure.
Time Frame: From "anesthesia start" to "anesthesia end", on average 5 hours
Measure: Mean (Standard Deviation); unit: bpm
Arm/Group | LMA Gastro | Standard of Care
Number analyzed (Participants) | 26 | 30
bpm
  Heart rate prior to intervention | 79.8846 (16.7412) | 77.3667 (13.7853)
  Heart rate post intervention | 77.1154 (15.8501) | 66.9667 (10.3607)

8. Secondary Outcome: To Describe Blood Pressure and End Tidal Carbon Dioxide [CO2] Within the Two Groups
Description: Blood pressure and end tidal carbon dioxide [CO2] were measured prior treatment administration and at the end of the procedure.
Time Frame: From "anesthesia start" to "anesthesia end", on average 5 hours
Measure: Mean (Standard Deviation); unit: mmhg
Arm/Group | LMA Gastro | Standard of Care
Number analyzed (Participants) | 26 | 30
mmhg
  Systolic Blood pressure prior to intervention | 127.2308 (19.4757) | 137.5714 (28.3097)
  Systolic Blood pressure post intervention | 122.0769 (15.0676) | 128.2 (23.5231)
  Diastolic Blood pressure prior to intervention | 78.3462 (10.7664) | 80.8571 (15.1846)
  Diastolic Blood pressure post intervention | 76.9231 (10.0833) | 77.7 (15.0611)
  End tidal carbon dioxide [CO2] prior to intervention | 18.6364 (11.4129) | 25.2 (11.7858)
  End tidal carbon dioxide [CO2] post intervention | 22.0769 (9.1693) | 28.75 (10.707)

9. Secondary Outcome: To Describe Oxygen Saturations Within the Two Groups
Description: Oxygen saturations were measured prior treatment administration and at the end of the procedure.
Time Frame: From "anesthesia start" to "anesthesia end", on average 5 hours
Measure: Mean (Standard Deviation); unit: percentage of saturation
Arm/Group | LMA Gastro | Standard of Care
Number analyzed (Participants) | 26 | 30
percentage of saturation
  Oxygen saturation prior to intervention | 98.5769 (1.9426) | 99.033 (1.1885)
  Oxygen saturation post intervention | 93.7692 (1.6796) | 98.5 (1.9783)

10. Secondary Outcome: To Evaluate Anesthesiologist Placing the Device
Description: Number of attempts means how many times the anesthesiologist tried to secure airway.
Time Frame: At the end of procedure, between 5 - 10 minutes
Population: This outcome is evaluating the providers not participants. This outcome is only applicable to the LMA Gastro arm since it is in this arm we are using the study device.
Measure: Number; unit: percentage of successful attempts
Arm/Group | LMA Gastro | Standard of Care
Number analyzed (Participants) | 5 | 0
percentage of successful attempts
  Successful on Attempt 1 | 77 |
  Successful on Attempt 2 | 19 |
  Successful on Attempt 3 | 4 |

ADVERSE EVENTS:
Time Frame: Since anesthesia start to discharge ready in PACU, up to 5 hours
Arm/Group | LMA Gastro | Standard of Care
All-Cause Mortality (participants affected / at risk) | 0/26 | 0/30
Serious Adverse Events (participants affected / at risk) | 0/26 | 0/30
Other Adverse Events (participants affected / at risk) | 24/26 | 3/30
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | LMA Gastro (N=26) | Standard of Care (N=30)
Horseness (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 1 (1)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 13 (13) | 2 (2)
Sore mouth (General disorders) | 2 (2) | 0 (0)
Sore Jaw (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Dysphagia (General disorders) | 4 (4) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-06-23): https://cdn.clinicaltrials.gov/large-docs/64/NCT04740164/Prot_SAP_001.pdf